CLINICAL TRIAL: NCT05438602
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 2, RANDOMIZED, DOUBLE-BLIND, 3-ARM STUDY TO INVESTIGATE NIRMATRELVIR/RITONAVIR IN NONHOSPITALIZED PARTICIPANTS AT LEAST 12 YEARS OF AGE WITH SYMPTOMATIC COVID-19 WHO ARE IMMUNOCOMPROMISED
Brief Title: A Study to Learn About the Study Medicines (Nirmatrelvir Plus Ritonavir) in People Aged 12 Years or Older With COVID-19 and a Compromised Immune System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C4671034; 2022-001362-35 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-06-30 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Coronavirus disease 2019 (COVID-19); Paxlovid; Nirmatrelvir; Immunocompromised
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nirmatrelvir plus ritonavir for 5 days (Experimental): Nirmatrelvir (2 tablets) plus ritonavir (1 capsule) will be given by mouth every 12 hours for 5 days followed by placebo for nirmatrelvir (2 tablets) plus placebo for ritonavir (1 capsule) every 12 hours for 10 days
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir; Drug: Placebo for nirmatrelvir; Drug: Placebo for ritonavir
- Nirmatrelvir plus ritonavir for 10 days (Experimental): Nirmatrelvir (2 tablets) plus ritonavir (1 capsule) will be given by mouth every 12 hours for 10 days followed by placebo for nirmatrelvir (2 tablets) plus placebo for ritonavir (1 capsule) every 12 hours for 5 days
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir; Drug: Placebo for nirmatrelvir; Drug: Placebo for ritonavir
- Nirmatrelvir plus ritonavir for 15 days (Experimental): Nirmatrelvir (2 tablets) plus ritonavir (1 capsule) will be given by mouth every 12 hours for 15 days.
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir — Participants will receive 2 tablets of nirmatrelvir every 12 hours
Drug: Ritonavir — Participants will receive 1 capsule of ritonavir every 12 hours
Drug: Placebo for nirmatrelvir — Participants will receive 2 tablets of placebo for nirmatrelvir every 12 hours. A placebo does not have any medicine in it but looks just like the medicine being studied.
  Arms: Nirmatrelvir plus ritonavir for 10 days; Nirmatrelvir plus ritonavir for 5 days
Drug: Placebo for ritonavir — Participants will receive 1 capsule of placebo for ritonavir every 12 hours. A placebo does not have any medicine in it but looks just like the medicine being studied.
  Arms: Nirmatrelvir plus ritonavir for 10 days; Nirmatrelvir plus ritonavir for 5 days

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called Nirmatrelvir/Ritonavir) for the possible treatment of COVID-19.

Patients with COVID-19 who have more difficulty in fighting against infections have a higher chance of severe illness. Such patients may benefit from longer treatment durations compared to the standard treatment regimen.

The study is seeking participants who:

* Have a confirmed COVID-19 infection
* Are Immunocompromised
* Experience onset of signs/symptoms attributable to the current COVID-19 infection within 5 days prior to screening and ≥1 signs/symptoms attributable to COVID-19 present on the day of randomization.

In addition, this study will also evaluate the efficacy and safety of a second treatment course of nirmatrelvir/ritonavir in people who experience that their COVID-19 is flaring up within 14 days of having taken a 5-day treatment course of nirmatrelvir/ritonavir.

For this group, the study is seeking participants who:

* Have a confirmed COVID-19 infection
* Experience a worsening of signs/symptoms after completing an initial 5-day course of nirmatrelvir/ritonavir
* The worsening of COVID-19 symptoms must occur within 14 days after completion of the initial 5-day course of nirmatrelvir/ritonavir
* Are Immunocompromised
* Experience onset of signs/symptoms attributable to the current COVID-19 infection within 48 hours prior to screening and ≥1 signs/symptoms attributable to COVID-19 present on the day of randomization.

All participants will be taking the study medicine for either 5, 10, or 15 days. The study medication will be taken by mouth 2 times a day. Participants will take part in this study for about 24 weeks. The first dose of study medication is taken at the study site and the rest at home. Selected participants will need to visit the study site at least 10 times during the study.

ELIGIBILITY:
Inclusion Criteria (applicable for both the main population and population with rebound):

* Participants aged 12 years or older and weighing ≥40 kg at screening.
* Immunocompromised
* ≥1 signs/symptoms attributable to COVID-19 present on the day of randomization.

Participants for the main population must have:

- Confirmed SARS-CoV-2 infection as determined by RT-PCR or other acceptable test method in any specimen collected within 5 days prior to randomization for the main study population.

Participants form the rebound population must have:

- Confirmed SARS-CoV-2 infection as determined by RT-PCR or rapid antigen testing in any specimen collected within 24h prior to randomization and collected within 14 days after the completion of the initial 5-day treatment course of nirmatrelvir/ritonavir for the population with rebound.

Exclusion Criteria:

* Current need for hospitalization or anticipated need for hospitalization within 24 h after randomization
* Known medical history of active liver disease
* Known HIV infection with a viral load >400 copies/mL or taking prohibited medications for human immunodeficiency virus (HIV)
* Receiving dialysis or have known age-specific estimated glomerular filtration rate (eGFR) or estimated creatinine clearance (eCrCl) <30 mL/min/1.73 m2 at screening as measured by a serum creatinine point of care device
* Oxygen saturation of <92% on room air obtained at rest within 24 hours prior to randomization
* Current use of any prohibited concomitant medication(s)
* Females who are pregnant and <14 weeks gestation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (25):
  - CRS Outpatient Services UCSF, San Francisco, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - UCSf infectious disease Lab, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - I.V.A.M. Clinical & Investigational Center, Doral, Florida
  - Qway Research LLC, Hialeah, Florida
  - Premium Medical Research Corp, Miami, Florida
  - Global Health Clinical Trials, Miami, Florida
  - I.V.A.M. Clinical & Investigational Center, Miami, Florida
  - NAPA Research, Pompano Beach, Florida
  - Santos Research Center, Tampa, Florida
  - Emory University Hospital-Georgia Clinical Research Center, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - National Institute of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont Infectious Diseases Research, Royal Oak, Michigan
  - Revival Research Institute, Sterling Heights, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - South Texas Clinical Research, Corpus Christi, Texas
  - Baylor University Medical Center, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A, Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - Fred Hutchinson Cancer Center - COVID Clinical Research Center, Seattle, Washington
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Royal Melbourne Hospital - Royal Park Campus, Parkville, Victoria
- Brazil (5):
  - Centro de Estudos e Pesquisa em Molestias Infecciosas - CPCLIN/RN, Natal, Rio Grande do Norte
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro
- Bulgaria (7):
  - Diagnostic Consultative Center - 1 Lom EOOD, Lom, Montana
  - MHAT Samokov, Samokov, Sofia
  - Military Medical Academy, Sofia, Sofia (stolitsa)
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases - Haskovo EOOD, Haskovo
  - MHAT - Heart and Brain, Pleven
  - Medical Center Artmed, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
- Canada (9):
  - Vancouver Infectious Diseases Centre, Vancouver, British Columbia
  - Dawson Clinical Research, Guelph, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - INTERMED Groupe Sante, Chicoutimi, Quebec
  - Clinique Medicale lActuel, Montreal, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Trois-Rivieres Inc., Sherbrooke, Quebec
- Hungary (3):
  - Medifarma 98 Kft, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Dél-Pesti Centrumkórház Országos Hematológiai és infektológiai intézet, Szent László telep, Budapest
  - Semmelweis Egyetem, Budapest
- Mexico (7):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - EME RED Hospitalaria, Mérida, Yucatán
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
  - FAICIC S. de R.L. de C.V., Veracruz
- Slovakia (12):
  - REUMEX s.r.o., Rimavská Sobota, Banská Bystrica Region
  - Narodny onkologicky ustav, Bratislava, Bratislava Region
  - ALERGIA s.r.o., Topoľčany, Nitra Region
  - MUDr. Viliam Cibik, PhD., s.r.o., Pruské, Trenčín Region
  - Univerzitna nemocnica Bratislava - Nemocnica sv. Cyrila a Metoda, Bratislava
  - Univerzitná nemocnica Bratislava, Nemocnica sv. Cyrila a Metoda, Bratislava
  - ARTROMAC n. o., Košice
  - MEDIKOMP, s.r.o, Prešov
  - Plucna ambulancia Hrebenar s.r.o., Spišská Nová Ves
  - Plucna ambulancia Hrebenar, s.r.o., Spišská Nová Ves
  - SANARE spol.s.r.o., Svidník
  - ALERGIA s.r.o., Topoľčany
- Spain (13):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra [pontevedra]
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mokgokong R, Cislo P, Tudone E, Weinstein E, Cappelleri JC. Symptom Alleviation/Resolution and Returns to Usual Health/Activities in Immunocompromised Adults with COVID-19 Treated with Nirmatrelvir-Ritonavir: Results from the EPIC-IC Trial. Infect Dis Ther. 2025 Dec;14(12):2763-2783. doi: 10.1007/s40121-025-01228-w. Epub 2025 Oct 14. PMID 41085942
- [Derived] Weinstein E, Paredes R, Gardner A, Almas M, Baniecki ML, Guan S, Tudone E, Antonucci S, Gregg K, Garcia-Vidal C, Camacho-Ortiz A, Wisemandle W, Terra SG, Liu S, Aberg JA, Rana MM, Corey L, Ford ES, Hammond J, Rusnak J. Extended nirmatrelvir-ritonavir treatment durations for immunocompromised patients with COVID-19 (EPIC-IC): a placebo-controlled, randomised, double-blind, phase 2 trial. Lancet Infect Dis. 2025 Nov;25(11):1243-1253. doi: 10.1016/S1473-3099(25)00221-X. Epub 2025 Jul 14. PMID 40675169
- [Derived] Baniecki ML, Guan S, Rai DK, Yang Q, Lee JT, Hao L, Weinstein E, Hyde C, Cardin RD, Soares H, Hammond J. Integrated virologic analysis of resistance to nirmatrelvir/ritonavir in individuals across four phase 2/3 clinical studies for the treatment of COVID-19. EBioMedicine. 2025 Aug;118:105819. doi: 10.1016/j.ebiom.2025.105819. Epub 2025 Jun 30. PMID 40592258
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study there were following population enrolled: main study population (MSP) and rebound population (RP). MSP: Non-hospitalized participants aged greater than or equal to (>=) 12 years weighing >= 40 kilogram(kg) who were immunocompromised and diagnosed with symptomatic Coronavirus disease 2019 (COVID-19) were enrolled. RP: Non-hospitalized participants with documented, symptomatic COVID-19 rebound within 14 days after 5-day treatment with nirmatrelvir/ritonavir were enrolled.
Groups:
- Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day: Eligible participants were randomized to receive nirmatrelvir 300 milligram (mg) and ritonavir 100 mg orally every 12 hours (q12h) for 5 days. Participants with estimated glomerular filtration rate (eGFR) >=30 to less than (<) 60 milliliters per minute (mL/min)/1.73 square meter (m^2) or estimated creatinine clearance (eCrCl) >=30 to <60 mL/min received nirmatrelvir 150 mg and ritonavir 100 mg orally q12h for 5 days. Participants then received placebo for nirmatrelvir and placebo for ritonavir q12h for next 10 days. Participants had follow-up through Day 44. Participants had long term follow-up through Week 24.
- Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day: Eligible participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally q12h for 10 days. Participants with eGFR >=30 to <60 mL/min/1.73 m^2 or eCrCl >=30 to <60 mL/min received nirmatrelvir 150 mg and ritonavir 100 mg orally q12h for 10 days. Participants then received placebo for nirmatrelvir and placebo for ritonavir q12h for next 5 days. Participants had follow-up through Day 44. Participants had long term follow-up through Week 24.
- Nirmatrelvir + Ritonavir 15 Day: Eligible participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally q12h for 5 days. Participants with eGFR >=30 to <60 mL/min/1.73 m^2 or eCrCl >=30 to <60 mL/min received nirmatrelvir 150 mg and ritonavir 100 mg orally q12h for 15 days. Participants had follow-up through Day 44. Participants had long term follow-up through Week 24.
Period: Treatment (15 Days)
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Started | 54 | 52 | 51
Completed | 50 | 49 | 43
Not Completed | 4 | 3 | 8
Not completed — Adverse Event | 2 | 1 | 3
Not completed — No longer met eligibility criteria | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 4
Period: Follow-up (Through Day 44)
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Started | 54 (Participants followed up after discontinuation or completion of treatment.) | 52 (Participants followed up after discontinuation or completion of treatment.) | 51 (Participants followed up after discontinuation or completion of treatment.)
Completed | 50 | 50 | 45
Not Completed | 4 | 2 | 6
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 6
Period: Long-term Follow-up (Through Week 24)
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Started | 54 (Participants followed up after discontinuation or completion of treatment.) | 52 (Participants followed up after discontinuation or completion of treatment.) | 51 (Participants followed up after discontinuation or completion of treatment.)
Completed | 47 | 47 | 44
Not Completed | 7 | 5 | 7
Not completed — Other | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Safety population included all randomised participants who received at least 1 dose of the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day | Total
Number analyzed (Participants) | 54 | 52 | 51 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.09 (14.77) | 54.77 (16.20) | 55.63 (14.44) | 55.85 (15.08)
Age, Customized [Count of Participants; unit: Participants]
  < 12 years | 0 | 0 | 0 | 0
  12 - 17 years | 0 | 1 | 0 | 1
  18 - 44 years | 11 | 9 | 11 | 31
  45 - 59 years | 19 | 19 | 17 | 55
  60 - 64 years | 4 | 7 | 10 | 21
  65 - 74 years | 14 | 11 | 8 | 33
  >= 75 years | 6 | 5 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 26 | 84
  Male | 26 | 22 | 25 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 33 | 32 | 101
  Not Hispanic or Latino | 16 | 19 | 19 | 54
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 3 | 7
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 50 | 47 | 44 | 141
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Nasopharyngeal (NP) Swab Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Ribonucleic Acid (RNA) < Lower Limit of Quantitation (LLOQ) From Day 15 to Day 44
Description: NP swab was collected by healthcare professional (HCP) from participants and were sent to the central laboratory for viral RNA level testing real-time reverse transcriptase-polymerase chain reaction(RT-PCR). Sustained was defined as NP swab SARS-CoV-2 RNA level not >=2.0 log10 per milliliter (copies/mL) at any study visit (through Day 44) following the first study visit where the participant's NP swab SARS-CoV-2 RNA level <LLOQ (<2.0 log10 copies/mL).
Time Frame: From Day 15 to Day 44
Population: Evaluable analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants | 61.54 (0.483) [0.483 to 0.748] | 70.83 (0.580) [0.580 to 0.837] | 66.00 (0.529) [0.529 to 0.791]

2. Secondary Outcome: Time to First NP Swab SARS-Cov-2 RNA <LLOQ for Participants With NP Swab SARS-CoV-2 RNA >= LLOQ at Baseline
Description: An NP swab was collected by HCP from participants and were sent to the central laboratory for viral RNA level testing RT-PCR. The LLOQ is <2.0 log10 copies/mL. Kaplan-Meier method was used for analysis. Time (days) to first NP swab SARS-CoV-2 RNA<LLOQ (event) was calculated as (First Event Date) - (First Dose Date) +1.
Time Frame: Day 1 through Day 44
Population: Evaluable analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure with non-missing data in the analysis set.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 46 | 44 | 45
Days | 9.500 (6.000) [6.000 to 15.000] | 11.000 (10.000) [10.000 to 15.000] | 9.000 (6.000) [6.000 to 11.000]

3. Secondary Outcome: Time to First Sustained NP Swab SARS-CoV-2 RNA < LLOQ for Participants Through Day 44 With NP Swab SARS-CoV-2 RNA >= LLOQ at Baseline
Description: An NP swab was collected by HCP from participants and were sent to the central laboratory for viral RNA level testing RT-PCR. Sustained was defined as NP swab SARS-CoV-2 RNA level not >=2.0 log10 copies/mL at any study visit (through Day 44) following the first study visit where the participant's NP swab SARS-CoV-2 RNA level < LLOQ. The LLOQ is <2.0 log10 copies/mL. Time (days) to first sustained NP swab SARS-CoV-2 RNA<LLOQ (event) was calculated as (First Event Date) - (First Dose Date) +1.
Time Frame: Day 1 through Day 44
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 46 | 44 | 45
Days | 15.000 (9.000) [9.000 to 16.000] | 11.000 (10.000) [10.000 to 15.000] | 10.000 (9.000) [9.000 to 16.000]

4. Secondary Outcome: Percentage of Participants With SARS-CoV-2 RNA < LLOQ in Plasma Over Time at Each Visit Through Week 24
Description: A 6-mL blood sample was collected for adult and pediatric participants and was analyzed to measure SARS-CoV-2 RNA <LLOQ in Plasma by RT-PCR. The LLOQ is <2.0 log10 copies/mL.
Time Frame: Baseline; Days 5, 10, 15, 21, 28, 35, and 44; Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Baseline | 98.08 (0.930) [0.930 to 1.000] | 97.92 (0.925) [0.925 to 1.000] | 92.00 (0.923) [0.923 to 1.000]
  Day 5 | 90.38 (0.925) [0.925 to 1.000] | 93.75 (0.921) [0.921 to 1.000] | 92.00 (0.923) [0.923 to 1.000]
  Day 10 | 92.31 (0.926) [0.926 to 1.000] | 95.83 (0.923) [0.923 to 1.000] | 92.00 (0.923) [0.923 to 1.000]
  Day 15 | 88.46 (0.923) [0.923 to 1.000] | 91.67 (0.920) [0.920 to 1.000] | 88.00 (0.920) [0.920 to 1.000]
  Day 21 | 86.54 (0.921) [0.921 to 1.000] | 93.75 (0.921) [0.921 to 1.000] | 88.00 (0.920) [0.920 to 1.000]
  Day 28 | 84.62 (0.920) [0.920 to 1.000] | 95.83 (0.923) [0.923 to 1.000] | 78.00 (0.910) [0.910 to 1.000]
  Day 35 | 82.69 (0.918) [0.918 to 1.000] | 93.75 (0.921) [0.921 to 1.000] | 84.00 (0.916) [0.916 to 1.000]
  Day 44 | 86.54 (0.921) [0.921 to 1.000] | 91.67 (0.920) [0.920 to 1.000] | 88.00 (0.920) [0.920 to 1.000]
  Week 12 | 73.08 | 87.50 | 78.00
  Week 24 | 69.23 | 85.42 | 84.00

5. Secondary Outcome: Percentage of Participants With SARS-CoV-2 RNA <LLOQ in NP Swabs at Each Study Visit Through Day 44
Description: An NP swab was collected by HCP from adult and pediatric participants and were sent to the central laboratory for viral RNA level testing RT-PCR. The LLOQ is <2.0 log10 copies/mL.
Time Frame: Baseline; Days 5, 10, 15, 21, 28, 35 and 44
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Baseline | 5.77 (0.292) [0.292 to 1.000] | 8.33 (0.398) [0.398 to 1.000] | 4.00 (0.158) [0.158 to 1.000]
  Day 5 | 38.46 (0.832) [0.832 to 1.000] | 29.17 (0.768) [0.768 to 1.000] | 38.00 (0.824) [0.824 to 1.000]
  Day 10 | 51.92 (0.872) [0.872 to 1.000] | 64.58 (0.888) [0.888 to 1.000] | 58.00 (0.881) [0.881 to 1.000]
  Day 15 | 69.23 (0.903) [0.903 to 1.000] | 77.08 (0.905) [0.905 to 1.000] | 72.00 (0.903) [0.903 to 1.000]
  Day 21 | 71.15 (0.905) [0.905 to 1.000] | 91.67 (0.920) [0.920 to 1.000] | 78.00 (0.910) [0.910 to 1.000]
  Day 28 | 80.77 (0.916) [0.916 to 1.000] | 93.75 (0.921) [0.921 to 1.000] | 76.00 (0.907) [0.907 to 1.000]
  Day 35 | 80.77 (0.916) [0.916 to 1.000] | 91.67 (0.920) [0.920 to 1.000] | 84.00 (0.916) [0.916 to 1.000]
  Day 44 | 78.85 (0.914) [0.914 to 1.000] | 91.67 (0.920) [0.920 to 1.000] | 88.00 (0.920) [0.920 to 1.000]

6. Secondary Outcome: Change From Baseline in SARS-CoV-2 RNA Level in NP Swabs at Days 5, 10, 15, 21, 28, 35 and 44
Description: An NP swab was collected by HCP from adult and pediatric participants and were sent to the central laboratory for viral RNA level testing RT-PCR.
Time Frame: Baseline; Days 5, 10, 15, 21, 28, 35 and 44
Population: Evaluable analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Here "Number of Participants Analyzed" were participants evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to table but may not have evaluable data for every row. Here, "number analyzed" signifies participants with non-missing data in the analysis set and evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
log10 copies/mL
  Change at Day 5: number analyzed (Participants) | 45 | 43 | 45
  Change at Day 5 | -3.449 (1.730) | -3.621 (1.521) | -3.746 (1.687)
  Change at Day 10: number analyzed (Participants) | 45 | 43 | 45
  Change at Day 10 | -4.167 (2.292) | -4.931 (1.899) | -5.002 (1.942)
  Change at Day 15: number analyzed (Participants) | 44 | 42 | 42
  Change at Day 15 | -4.827 (2.476) | -5.773 (1.473) | -6.009 (2.093)
  Change at Day 21: number analyzed (Participants) | 42 | 42 | 40
  Change at Day 21 | -5.472 (2.028) | -6.328 (1.472) | -6.319 (1.967)
  Change at Day 28: number analyzed (Participants) | 43 | 42 | 38
  Change at Day 28 | -5.938 (2.138) | -6.509 (1.571) | -6.530 (1.770)
  Change at Day 35: number analyzed (Participants) | 40 | 41 | 42
  Change at Day 35 | -6.237 (1.746) | -6.596 (1.453) | -6.633 (1.816)
  Change at Day 44: number analyzed (Participants) | 42 | 42 | 42
  Change at Day 44 | -5.916 (1.865) | -6.597 (1.445) | -6.707 (1.922)

7. Secondary Outcome: Change From Baseline in SARS-CoV-2 RNA Level in Plasma at Days 5, 10, 15, 21, 28, 35 and 44
Description: A 6-mL blood sample was collected for adult and pediatric participants and was analyzed to measure SARS-CoV-2 RNA by RT-PCR.
Time Frame: Baseline; Days 5, 10, 15, 21, 28, 35 and 44
Population: Evaluable analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants with non-missing data in the analysis set and evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 8 | 10 | 15
log10 copies/mL
  Change at Day 5: number analyzed (Participants) | 7 | 10 | 15
  Change at Day 5 | -1.457 (0.643) | -1.360 (0.717) | -1.528 (0.626)
  Change at Day 10: number analyzed (Participants) | 8 | 9 | 14
  Change at Day 10 | -1.487 (0.601) | -1.700 (0.000) | -1.880 (0.380)
  Change at Day 15: number analyzed (Participants) | 8 | 9 | 14
  Change at Day 15 | -1.700 (0.000) | -1.700 (0.000) | -1.880 (0.380)
  Change at Day 21: number analyzed (Participants) | 7 | 10 | 14
  Change at Day 21 | -1.700 (0.000) | -1.700 (0.000) | -1.880 (0.380)
  Change at Day 28: number analyzed (Participants) | 7 | 10 | 12
  Change at Day 28 | -1.700 (0.000) | -1.700 (0.000) | -1.910 (0.405)
  Change at Day 35: number analyzed (Participants) | 7 | 10 | 13
  Change at Day 35 | -1.700 (0.000) | -1.700 (0.000) | -1.894 (0.392)
  Change at Day 44: number analyzed (Participants) | 7 | 10 | 14
  Change at Day 44 | -1.700 (0.000) | -1.700 (0.000) | -1.880 (0.380)

8. Secondary Outcome: Number of Participants With Rebound in SARS-CoV-2 RNA Level in NP Swabs at Follow up
Description: Rebound in SARS-CoV-2 RNA level in NP swabs at follow up (ie, any study visit after end of treatment through Day 44) was defined as a half (0.5) log10 copies/mL increase or greater in SARS-CoV-2 RNA level relative to end of treatment SARS-CoV-2 RNA level based on treatment regimen, with a follow-up viral RNA level >= 2.5 log10 copies/mL.
Time Frame: Day 16 through Day 44
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Participants | 9 | 1 | 1

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Treatment Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start emerges. SAE was an AE resulting in any of the following outcomes or considered medically significant: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or birth defect.
Time Frame: Day 1 of dosing up to Week 24
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 54 | 52 | 51
Participants
  TEAEs | 28 | 34 | 31
  SAEs | 5 | 1 | 4
  AEs Leading to Study Treatment Discontinuation | 1 | 1 | 4

10. Secondary Outcome: Percentage of Participants With COVID-19-Related Hospitalization >24 Hours (h) or Death Through Day 28
Description: Hospitalization >24 h is defined as >24h of acute care in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with severe COVID-19. This included specialized acute medical care unit within an assisted living facility or nursing home. This did not include hospitalization for the purposes of public health and/or clinical trial execution.
Time Frame: Day 1 through Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Hospitalization | 3.846 | 0 | 0
  Death | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Death Through Week 24
Description: Death due to any cause through week 24 was considered. Kaplan-Meier method was used for evaluation.
Time Frame: Day 1 through Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants | 1.923 | 0 | 0

12. Secondary Outcome: Percentage of Participants With COVID-19-Related Hospitalization Through Day 44 and Week 24
Description: COVID-19 related hospitalization is defined as >24h of acute care in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with severe COVID-19. This included specialized acute medical care unit within an assisted living facility or nursing home. This did not include hospitalization for the purposes of public health and/or clinical trial execution.
Time Frame: Day 1 through Day 44 and Day 1 through Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Through Day 44 | 3.846 | 0 | 0
  Through Week 24 | 3.846 | 0 | 0

13. Secondary Outcome: Percentage of Participants With COVID-19-Related Intensive Care Unit (ICU) Admission Through Day 44 and Week 24
Time Frame: Day 1 through Day 44 and Day 1 through Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Through Day 44 | 1.923 | 0 | 0
  Through Week 24 | 1.923 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) Through Day 44 and Week 24
Description: Invasive mechanical ventilation or ECMO were types of oxygen support received in hospital.
Time Frame: Day 1 through Day 44 and Day 1 through Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants
  Through Day 44 | 0 | 0 | 0
  Through Week 24 | 0 | 0 | 0

15. Secondary Outcome: Mean Number of Days in Hospital and ICU Stay Through Day 44 and Through Week 24
Description: Hospitalization >24 hours is defined as >24h of acute care in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with severe COVID-19.
Time Frame: Day 1 through Day 44 and Day 1 through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Days
  Hospital Stay: Up to Day 44 | 0.635 (3.453) [lower limit 3.453] | 0.000 (0.000) [lower limit 0.000] | 0.000 (0.000) [lower limit 0.000]
  Hospital Stay: Up to Week 24 | 0.635 (3.453) [lower limit 3.453] | 0.000 (0.000) [lower limit 0.000] | 0.000 (0.000) [lower limit 0.000]
  ICU Stay: Up to Day 44 | 0.442 (3.190) [lower limit 3.190] | 0.000 (0.000) [lower limit 0.000] | 0.000 (0.000) [lower limit 0.000]
  ICU Stay: Up to Week 24 | 0.442 (3.190) [lower limit 3.190] | 0.000 (0.000) [lower limit 0.000] | 0.000 (0.000) [lower limit 0.000]

16. Secondary Outcome: Mean Number of COVID-19-Related Medical Visits Through Day 44 and Through Week 24
Time Frame: Day 1 through Day 44 and Day 1 through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Medical visits
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Medical visits
  Through Day 44 | 0.115 (0.615) [lower limit 0.615] | 0.000 (0.000) [lower limit 0.000] | 0.000 (0.000) [lower limit 0.000]
  Through Week 24 | 0.115 (0.615) [lower limit 0.615] | 0.000 (0.000) [lower limit 0.000] | 0.020 (0.141) [lower limit 0.141]

17. Secondary Outcome: Time to First Alleviation of Each Targeted Signs and Symptoms Through Day 44
Description: Symptoms alleviation through day44 of each targeted COVID-19 sign/symptom was defined as first time when each targeted symptom scored as moderate/severe at study entry are scored as mild or absent and a targeted symptom scored mild or absent at study entry are scored as absent.COVID-19 targeted signs/symptoms were muscle or body aches,shortness of breath(SOB)or difficulty breathing,chills or shivering, cough,diarrhea,feeling hot or feverish,headache,nausea,stuffy or runny nose,sense of smell,sense of taste,sore throat,low energy or tiredness, vomit.
Time Frame: Day 1 through Day 44
Population: Evaluable analysis set analyzed. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed"' contributed data to table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with non-missing data and with baseline severity of mild, moderate and severe of targeted signs/symptoms.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Days
  Muscle or body aches: number analyzed (Participants) | 36 | 39 | 41
  Muscle or body aches | 6.000 [4.000 to 9.000] | 9.000 [4.000 to 9.000] | 9.000 [5.000 to 13.000]
  SOB or difficulty breathing: number analyzed (Participants) | 26 | 32 | 26
  SOB or difficulty breathing | 6.000 [4.000 to 9.000] | 9.000 [4.000 to 9.000] | 6.000 [4.000 to 13.000]
  Chills or shivering: number analyzed (Participants) | 27 | 34 | 33
  Chills or shivering | 5.000 [4.000 to 6.000] | 4.000 [4.000 to 5.000] | 5.000 [4.000 to 5.000]
  Cough: number analyzed (Participants) | 50 | 44 | 44
  Cough | 6.000 [5.000 to 9.000] | 9.000 [6.000 to 9.000] | 10.000 [5.000 to 13.000]
  Diarrhea: number analyzed (Participants) | 22 | 12 | 14
  Diarrhea | 9.000 [5.000 to 10.000] | 5.000 [4.000 to 9.000] | 9.000 [4.000 to 22.000]
  Feeling hot or feverish: number analyzed (Participants) | 39 | 32 | 34
  Feeling hot or feverish | 5.000 [4.000 to 6.000] | 4.000 [4.000 to 5.000] | 5.000 [4.000 to 5.000]
  Headache: number analyzed (Participants) | 33 | 37 | 38
  Headache | 9.000 [4.000 to 15.000] | 5.000 [4.000 to 9.000] | 5.000 [4.000 to 9.000]
  Nausea: number analyzed (Participants) | 11 | 18 | 13
  Nausea | 9.000 [4.000 to 13.000] | 4.000 [4.000 to 5.000] | 6.000 [4.000 to 13.000]
  Stuffy or runny nose: number analyzed (Participants) | 46 | 46 | 47
  Stuffy or runny nose | 9.000 [6.000 to 11.000] | 9.000 [5.000 to 9.000] | 9.000 [5.000 to 10.000]
  Sense of smell: number analyzed (Participants) | 15 | 21 | 20
  Sense of smell | 9.000 [6.000 to 10.000] | 9.000 [4.000 to 10.000] | 9.000 [5.000 to 10.000]
  Sense of taste: number analyzed (Participants) | 15 | 18 | 24
  Sense of taste | 10.000 [5.000 to 10.000] | 9.000 [4.000 to 10.000] | 9.000 [6.000 to 13.000]
  Sore throat: number analyzed (Participants) | 33 | 38 | 37
  Sore throat | 6.000 [4.000 to 6.000] | 5.000 [4.000 to 9.000] | 5.000 [4.000 to 9.000]
  Low energy or tiredness: number analyzed (Participants) | 45 | 46 | 46
  Low energy or tiredness | 9.000 [6.000 to 13.000] | 9.000 [5.000 to 10.000] | 9.000 [5.000 to 14.000]
  Vomit: number analyzed (Participants) | 5 | 4 | 6
  Vomit | 6.000 [4.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event. | 4.000 [NA to NA] — The number of participants response in the participant's diary and participants with events available were not sufficient for calculation of the limits using Kaplan-Meier method | 4.500 [4.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event.

18. Secondary Outcome: Time to First Resolution of Each Targeted Signs and Symptoms Through Day 44
Description: Symptoms resolution through day 44 of each targeted COVID-19 sign/symptom was defined as the first time when each targeted symptom scored as mild, moderate or severe at study entry are scored as absent. COVID -19 targeted signs/symptoms were muscle or body aches, SOB or difficulty breathing, chills or shivering, cough, diarrhoea, feeling hot or feverish, headache, nausea, stuffy or runny nose, sense of smell, sense of taste, sore throat, low energy or tiredness, vomit.
Time Frame: Day 1 through Day 44
Population: Evaluable analysis set analyzed. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed"' contributed data to table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with non-missing data and with baseline severity of mild, moderate and severe of targeted signs and symptoms.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Days
  Muscle or body aches: number analyzed (Participants) | 36 | 39 | 41
  Muscle or body aches | 14.500 [10.000 to 19.000] | 11.000 [9.000 to 21.000] | 10.000 [6.000 to 20.000]
  SOB or difficulty breathing: number analyzed (Participants) | 26 | 32 | 26
  SOB or difficulty breathing | 9.000 [5.000 to 13.000] | 9.500 [9.000 to 19.000] | 12.000 [6.000 to 19.000]
  Chills or shivering: number analyzed (Participants) | 27 | 34 | 33
  Chills or shivering | 6.000 [4.000 to 9.000] | 4.000 [4.000 to 9.000] | 5.000 [4.000 to 6.000]
  Cough: number analyzed (Participants) | 50 | 44 | 44
  Cough | 13.000 [10.000 to 20.000] | 12.000 [9.000 to 21.000] | 19.500 [11.000 to 22.000]
  Diarrhea: number analyzed (Participants) | 22 | 12 | 14
  Diarrhea | 9.000 [6.000 to 10.000] | 9.000 [4.000 to 13.000] | 16.500 [4.000 to 26.000]
  Feeling hot or feverish: number analyzed (Participants) | 39 | 32 | 34
  Feeling hot or feverish | 9.000 [5.000 to 9.000] | 7.000 [4.000 to 9.000] | 5.000 [4.000 to 6.000]
  Headache: number analyzed (Participants) | 33 | 37 | 38
  Headache | 13.000 [9.000 to 15.000] | 10.000 [9.000 to 15.000] | 9.000 [5.000 to 11.000]
  Nausea: number analyzed (Participants) | 11 | 18 | 13
  Nausea | 9.000 [4.000 to 14.000] | 4.000 [4.000 to 9.000] | 9.000 [4.000 to 13.000]
  Stuffy or runny nose: number analyzed (Participants) | 46 | 46 | 47
  Stuffy or runny nose | 14.000 [10.000 to 22.000] | 13.000 [9.000 to 15.000] | 13.000 [9.000 to 16.000]
  Sense of smell: number analyzed (Participants) | 15 | 21 | 20
  Sense of smell | 10.000 [9.000 to 15.000] | 9.000 [5.000 to 11.000] | 9.000 [5.000 to 10.000]
  Sense of taste: number analyzed (Participants) | 15 | 18 | 24
  Sense of taste | 10.000 [9.000 to 14.000] | 10.500 [9.000 to 21.000] | 10.000 [6.000 to 13.000]
  Sore throat: number analyzed (Participants) | 33 | 38 | 37
  Sore throat | 9.000 [5.000 to 11.000] | 9.500 [9.000 to 13.000] | 9.000 [9.000 to 10.000]
  Low energy or tiredness: number analyzed (Participants) | 45 | 46 | 46
  Low energy or tiredness | 27.000 [13.000 to 33.000] | 20.000 [13.000 to 35.000] | 22.000 [15.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event.
  Vomit: number analyzed (Participants) | 5 | 4 | 6
  Vomit | 6.000 [4.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event. | 4.000 [4.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event. | 4.500 [4.000 to NA] — The upper limit of CI could not be estimated due to insufficient number of participants with event.

19. Secondary Outcome: Percentage of Participants With Any Severe Targeted Signs and Symptoms Attributed to COVID-19 Through Day 44
Description: COVID-19 targeted signs/symptoms were muscle or body aches, SOB or difficulty breathing, chills or shivering, cough, diarrhea, feeling hot or feverish, headache, nausea, stuffy or runny nose, sense of smell, sense of taste, sore throat, low energy or tiredness, vomit.
Time Frame: Day 1 through Day 44
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
Number analyzed (Participants) | 52 | 48 | 50
Percentage of participants | 28.85 | 31.25 | 38.00

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to Week 24
Description: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day | Nirmatrelvir + Ritonavir 15 Day
All-Cause Mortality (participants affected / at risk) | 1/54 | 0/52 | 1/51
Serious Adverse Events (participants affected / at risk) | 5/54 | 1/52 | 4/51
Other Adverse Events (participants affected / at risk) | 12/54 | 19/52 | 19/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day (N=54) | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day (N=52) | Nirmatrelvir + Ritonavir 15 Day (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day (N=54) | Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 Day (N=52) | Nirmatrelvir + Ritonavir 15 Day (N=51)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 6 (6) | 12 (12) | 14 (14)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
For outcome measure data have not been reported for RP separately, since there was 1 participant each in 2 arms (Nirmatrelvir + Ritonavir 5 Day Then Placebo 10 Day and Nirmatrelvir + Ritonavir 10 Day Then Placebo 5 day), it could have led to re-identification of RP participants. In other sections of results data for RP and MSP have been combined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT05438602/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT05438602/SAP_001.pdf